CLINICAL TRIAL: NCT02534844
Title: A Phase 2b/3 Prospective, Randomized, Double-Blind, Sham-Controlled 3-Part Trial of VTS-270 (2-hydroxypropyl-β-cyclodextrin) in Subjects With Neurologic Manifestations of Niemann-Pick Type C1 (NPC1) Disease
Brief Title: VTS-270 to Treat Niemann-Pick Type C1 (NPC1) Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mandos LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTS301 (Parts A/B); 2015-002548-15 (EudraCT Number)
Record Dates: First submitted 2015-08-18; First posted 2015-08-28 (Estimated); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Niemann-Pick Type C1 (NPC1) Disease; neurologic disease; gross motor dysfunction; fine motor dysfunction; dysphagia; swallowing problems; cognitive dysfunction; gait abnormalities; pediatrics
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Disease; Deglutition Disorders; Cognitive Dysfunction; Mobility Limitation | interventions — Cyclodextrins; 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Intervention Model Description: In Parts A/B (see other registration for Part C description)
Who Masked: Care Provider, Investigator
Masking Description: While it is a double-blind trial, the participant and outcomes assessor will be blinded, as well as the Care Provider and Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parts A/B: Sham Control (Experimental): Participants receive no study drug
  Interventions: Other: Parts A/B: Sham Control
- Parts A/B: Adrabetadex (Other): Participants receive adrabetadex
  Interventions: Drug: Parts A/B: Adrabetadex

INTERVENTIONS:
Drug: Parts A/B: Adrabetadex — 900 - 1800 milligram (mg) of adrabetadex administered every 2 weeks via lumbar intrathecal infusion
  Other Names: 2-hydroxypropyl-β-cyclodextrin; Cyclodextrin; VTS-270; Adrabetadex
  Arms: Parts A/B: Adrabetadex
Other: Parts A/B: Sham Control — No experimental drug is administered to participants - intrathecal administrations are simulated by skin prick
  Other Names: Procedure Control; Skin prick
  Arms: Parts A/B: Sham Control

SUMMARY:
Due to different study designs, the sponsor separated Part C into a separate registration (NCT04958642), leaving Parts A/B here in NCT02534844.

This study is to find out how safe and effective VTS-270 is for patients with Niemann-Pick Type C1 (NPC1) disease who have neurologic symptoms (listed under Keywords).

In Parts A/B, two out of every three patients will receive the study drug. The third patient will receive 1 to 2 small needle pricks at the location where the LP and IT injection is normally made (sham control).

In Part C, all participants will receive study drug, as described in the Part C registration record.

Start date for this record is the first day a participant was enrolled in Parts A/B. The trial is actually continuing until the last primary outcome measure of safety data are collected from Part C participants. The last primary outcome measure of safety, along with final adverse events results will be posted in the separate Part C registration record.

DETAILED DESCRIPTION:
Non-clinical studies and a Phase 1 clinical trial suggest that intrathecal administration of VTS-270 in patients with neurologic manifestations of Niemann-Pick Type C1 (NPC1) disease has the potential to slow the rate of progression of their neurologic disease.

Niemann-Pick Type C1 (NPC1) disease is a rare, neurodegenerative, inherited, autosomal recessive lysosomal lipid storage disorder primarily in children and teenagers. The disease is characterized by the inability to properly metabolize cholesterol and other lipids within the cell due to mutations in the NPC1 gene, causing unesterified cholesterol to accumulate in the brain, liver and spleen.

This study plans to enroll about 51 participants with NPC1 disease. It will be conducted in three parts: Parts A, B, and C.

* Part A will evaluate 3 different dose levels of VTS-270 in 12 participants to determine the dose level for Parts B and C.
* In Part B, 39 more participants will join the original 12 to evaluate the safety and effectiveness of the dose selected from Part A compared to sham control.
* Part C will be an open-label extension phase of the study for Part B participants who either complete Part B or have met rescue therapy criteria, as well as participants entering Part C from other trials.

Participants in Part C will receive treatment with VTS-270 until the product is licensed or the program is terminated (anticipated within 5 years).

Final results will be posted in the Part C registration record (NCT04958642).

ELIGIBILITY:
Key Inclusion Criteria:

Parts A/B:

1. Had onset of neurological symptoms prior to 15 years of age
2. Has confirmed diagnosis of NPC1 determined by either:

   1. two NPC1 mutations
   2. positive filipin staining and at least one NPC1 mutation
   3. vertical supranuclear gaze palsy (VSNGP) in combination with either: one NPC1 mutation, OR positive filipin staining or oxysterol levels consistent with NPC disease and no Niemann-Pick Type C2 (NPC2) Disease mutations
3. Adult participant or parent/guardian has provided written informed consent, with assent collected from minors of appropriate age
4. Is able to undergo a lumbar puncture (LP) and IT drug administration under conscious sedation or general anesthesia
5. Has an NPC Clinical Severity Scale Score of 1 through 4, inclusive, in two or more of the following components: ambulation, fine motor skills, or swallowing; and has a score of 0 through 4 on the cognition component
6. Has a total NPC Clinical Severity Scale Score of 10 or greater
7. If taking miglustat, must have been on a stable dose for past 6-8 weeks and be willing to remain on a stable dose
8. If participant has seizures, they have been adequately controlled for 3 months without changing dose or regimen
9. Has agreed to discontinue all non-prescription supplements at least 1 month prior to first dose (Study Day 0)
10. Has agreed to discontinue any other investigational treatments for NPC including vorinostat or arimoclomol at least 3 months prior to first dose (Study Day 0)
11. If of child-bearing potential (not surgically sterile), agrees to use a medically acceptable method continuously, until at least 30 days after participation in the study

Key Exclusion Criteria:

1. Has exclusion criteria as assessed by NPC Clinical Severity Scale:

   1. Unable to walk, wheelchair dependent (ambulation NPC score=5)
   2. Has need for a nasogastric tube to overcome swallowing difficulties (swallowing NPC score=5) unless used for supplemental feeding or administering medication
   3. severe dysmetria (fine motor score =5) or
   4. minimal cognitive function (cognition NPC score=5)
2. Weighs less than 15 kg
3. Has had prior treatment with intravenous 2-hydroxypropyl-β-cyclodextrin (HP-β-CD) for NPC1 disease, unless the subject has undergone a minimum 3-month washout period prior to Study Day 0, or has had any prior intrathecal (IT) administration of HP-β-CD
4. Is taking antipsychotics for treatment of psychosis; use of antipsychotic medication for treatment of other disorders (e.g., Attention Deficit Hyperactivity Disorder) will not exclude participation in this trial
5. Has a history of hypersensitivity reactions to any product containing HP-β-CD
6. Has a spinal deformity that could impact the ability to perform a lumbar puncture
7. Has had a skin infection in the lumbar region within 2 months of study entry
8. Has neutropenia, defined as an absolute neutrophil count (ANC) of less than 1.5 X 10^9/L
9. Has thrombocytopenia (platelet count of less than 75 X 10^9/L)
10. Has activated partial thromboplastin time (aPTT) or prothrombin time (PT) prolonged by > 1.5 times the upper limit of normal (ULN) or known history of a bleeding disorder
11. Has had status epilepticus occurring within 3 months of screening and/or seizure frequency that cannot be quantified
12. Has evidence of either obstructive hydrocephalus or normal pressure hydrocephalus
13. Has recently used anticoagulants [in past 2 weeks prior to first dose (Study Day 0); re: lumbar puncture safety].
14. Is unable to comply with the study procedures or has a clinical disease or laboratory abnormality that in the opinion of the investigator would potentially increase the risk of participation

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Lead, Study Director — Mandos LLC
Locations (29):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Shands Children's Hospital, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Eunice Kennedy Shriver National Institute of Child Health and Human Development, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Multicare Institute for Research and Innovation, Tacoma, Washington
- Australia (4):
  - The Prince of Wales Hospital, Sydney, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- CHU Paris Est - Hospital d'Enfants Armand-Trousseau, Paris, Cedex 12, France
- Germany (3):
  - Katholisches Klinikim Bochum gGmbH, Bochum
  - Universitaetsklinikum Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
- Waikato Hospital, Hamilton West, New Zealand
- National University Hospital (Singapore) Pte, Ltd, Singapore, Singapore
- Hospital Universitario del Valle Hebron, Barcelona, Spain
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Altındağ, Ankara
  - Gazi University Medical Faculty, Çankaya, Ankara
- United Kingdom (2):
  - Birmingham Women's and Children's NHS Trust, Birmingham, West Midlands
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: No
Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT02534844) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Farmer C, Lewis M, Farhat N, Robbins KP, Joseph L, Albert OK, Bianconi S, Hoffmann A, Giserman-Kiss I, Alexander DM, Thurm A, Porter FD, Kravis EB. Convergent Validity of the Fine Motor, Speech, and Cognitive Domains of the 5-Domain Niemann-Pick Disease Type C Clinical Severity Scale. J Child Neurol. 2026 Jan;41(1):43-53. doi: 10.1177/08830738251346348. Epub 2025 Jun 17. PMID 40525490

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Adrabetadex 900 mg: Participants received 4 lumbar intrathecal (IT) infusions of adrabetadex 900 milligrams (mg) once every 2 weeks.
- Part A: Adrabetadex 1200 mg: Participants received 4 lumbar IT infusions of adrabetadex 1200 mg once every 2 weeks.
- Part A: Adrabetadex 1800 mg: Participants received 4 lumbar IT infusions of adrabetadex 1800 mg once every 2 weeks.
- Part A: Sham Control; Part B: Sham Control: Participants received sham control procedures once every 2 weeks.
- Part B: Adrabetadex 900 mg: Participants received lumbar IT infusions of adrabetadex 900 mg once every 2 weeks.
Period: Part A
Arm/Group | Part A: Adrabetadex 900 mg | Part A: Adrabetadex 1200 mg | Part A: Adrabetadex 1800 mg | Part A: Sham Control | Part B: Adrabetadex 900 mg | Part B: Sham Control
Started | 3 | 3 | 3 | 3 | 0 | 0
Received at Least One Dose of Study Drug | 3 | 3 | 3 | 3 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Adrabetadex 900 mg | Part A: Adrabetadex 1200 mg | Part A: Adrabetadex 1800 mg | Part A: Sham Control | Part B: Adrabetadex 900 mg | Part B: Sham Control
Started | 0 | 0 | 0 | 0 | 29 | 15
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 29 | 15
Completed | 0 | 0 | 0 | 0 | 27 | 14
Not Completed | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population was defined as all randomized participants. As per planned analysis, baseline characteristics data were collected and presented by participants' overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study.
Groups:
- Sham Control: Participants received sham control procedures once every 2 weeks for a total of 52 weeks.
- Adrabetadex: Participants received lumbar IT infusions of adrabetadex once every 2 weeks for a total of 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Sham Control | Adrabetadex | Total
Number analyzed (Participants) | 18 | 38 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (5.10) | 12.7 (5.64) | 12.4 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 8 | 22 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 15 | 31 | 46
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 31 | 47
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Parts A/B: Change From Baseline to Week 52 in 4-Item Composite Score of Niemann Pick Type C Severity Scale (NPC-SS) Score
Description: The NPC-SS composite score is the sum of the ambulation, cognition, fine motor, and swallowing domains of the NPC-SS. Each of the four NPC-SS components (ambulation, cognition, fine motor, and swallowing) are rated on a scale from 0 (better) to 5 (worse). The total score was the sum of individual components scores which ranges from 0 (best) to 20 (worst), with higher scores indicating more severe clinical impairment.
Time Frame: Baseline, Week 52
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least one treatment (sham or adrabetadex). As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study. Here, number analyzed = participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
score on a scale
  Baseline: number analyzed (Participants) | 18 | 36
  Baseline | 8.1 (4.27) | 8.8 (3.12)
  Change from Baseline at Week 52 | -0.1 (1.55) | 0.0 (2.45)

2. Primary Outcome: Parts A/B: Number of Participants Classified With Each Score on the Clinician Global Impression of Change (CGIC) at Week 52
Description: The Clinician CGIC is a 7-point Likert scale. The scale requires assessment of change from a baseline level of disease activity, with anchors ranging from markedly improved, moderately improved, and minimally improved to no change and corresponding worsening (minimally, moderately, markedly). The Investigator rates his/her impression of the change in each participant's condition at week 52 on a scale from marked improvement (1) to marked worsening (7).
Time Frame: Week 52
Population: mITT population included all randomized participants who received at least one treatment (sham or adrabetadex). As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
Participants
  Markedly improved (1) | 0 | 0
  Moderately improved (2) | 1 | 5
  Minimally improved (3) | 4 | 9
  Unchanged (4) | 9 | 16
  Minimally worse (5) | 2 | 6
  Moderately worse (6) | 2 | 1
  Markedly worse (7) | 0 | 1

3. Secondary Outcome: Parts A/B: Change From Baseline to Week 52 in NPC-SS Total Score (Excluding Hearing and Auditory Brainstem Response [ABR])
Description: The NPC-SS total score is based on 9 domains including ambulation, fine motor skills, cognition, swallowing, memory, speech, eye movement, hearing (sensorineural) and seizures. The hearing domain and auditory brainstem response modifiers are removed from the total NPC-SS total score for this measure. A Likert-like scale is used to assign the remaining 8 major domain scores of 0 to 5 (better to worse). The total score was the sum of individual component scores which ranges from 0 (best) to 40 (worst), with higher scores indicating more severe clinical impairment.
Time Frame: Baseline, Week 52
Population: mITT population included all randomized participants who received at least one treatment. As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study. Here, overall number of participants analyzed = participants evaluable for this outcome measure. Number analyzed = participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 37
score on a scale
  Baseline | 16.94 (8.164) | 17.81 (6.476)
  Change from Baseline at Week 52 | -0.74 (2.357) | -0.34 (4.226)

4. Secondary Outcome: Parts A/ B: Number of Participants Classified as CGIC Responders at Week 52
Description: The Clinician CGIC is a 7-point Likert scale. The scale requires assessment of change from a baseline level of disease activity, with anchors ranging from markedly improved, moderately improved, and minimally improved to no change and corresponding worsening (minimally, moderately, markedly). The Investigator rates his/her impression of the change in each participant's condition at week 52 on a scale from marked improvement (1) to marked worsening (7). CGIC Responders are defined as participants who received the caregiver's rating of no change, minimally improved, moderately improved, or markedly improved from baseline to Week 52.
Time Frame: Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
Participants | 7 | 23

5. Secondary Outcome: Parts A/B: Number of Participants Classified as Responders on NPC-SS Total Score (Excluding Hearing and ABR) at Week 52
Description: The NPC-SS total score is based on 9 domains including ambulation, fine motor skills, cognition, swallowing, memory, speech, eye movement, hearing (sensorineural) and seizures. The hearing domain and ABR modifiers are removed from the total NPC-SS total score for this measure. A Likert-like scale is used to assign the remaining 8 major domain scores of 0 to 5 (better to worse). The total score was the sum of individual components scores which ranges from 0 (best) to 40 (worst), with higher scores indicating more severe clinical impairment. Responders on NPC-SS Total Score are defined as participants with no change or improvement on NPC-SS total score from baseline to Week 52.
Time Frame: Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
Participants | 13 | 22

6. Secondary Outcome: Parts A/B: EQ-5D-3L Questionnaire Visual Analog Scale (VAS) Score (for Health Status) at Baseline and at Week 52
Description: The EQ-5D-3L assessment is a self-reported, simple, descriptive system measuring 5 dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A vertical VAS allows the participants to indicate their health state that day, and ranges from 0 (worst imaginable) to 100 (best imaginable), with higher scores indicating better health state.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 37
score on a scale
  Baseline | 71.9 (16.28) | 68.3 (19.97)
  Week 52: number analyzed (Participants) | 15 | 34
  Week 52 | 73.2 (13.04) | 75.7 (19.00)

7. Secondary Outcome: Parts A/B: Number of Participants Treated for at Least 6 Months Who Qualified for the Rescue Option
Description: Participants who manifested significant disease progression according to predefined clinical criteria after treatment of 26 weeks or more had the option to rescue. Number of participants who qualified for the rescue option following a minimum of 26 weeks of treatment were analyzed.
Time Frame: Baseline up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
Participants | 2 | 2

8. Secondary Outcome: Parts A/B: Change From Baseline to Week 52 in Each of the 9 Clinical Domains of the NPC-SS
Description: The NPC-SS total score is based on 9 domains including ambulation, fine motor skills, cognition, swallowing, memory, speech, eye movement, hearing (sensorineural) and seizures. A Likert-like scale is used to assign to each domain score of 0 to 5 (better to worse) with higher scores indicating more severe clinical impairment.
Time Frame: Baseline, Week 52
Population: mITT population included all randomized participants who received at least one treatment (sham or adrabetadex). As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study. Here, Number analyzed = participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
score on a scale
  Ambulation (Baseline) | 1.83 (1.150) | 2.21 (1.298)
  Ambulation (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Ambulation (Change from Baseline at Week 52) | 0.00 (0.679) | 0.06 (1.434)
  Fine Motor (Baseline) | 2.06 (1.349) | 2.16 (1.128)
  Fine Motor (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Fine Motor (Change from Baseline at Week 52) | 0.07 (0.917) | 0.24 (1.103)
  Cognition (Baseline) | 2.56 (1.199) | 2.58 (1.222)
  Cognition (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Cognition (Change from Baseline at Week 52) | -0.14 (0.663) | 0.06 (0.919)
  Swallowing (Baseline) | 1.67 (1.495) | 1.79 (1.398)
  Swallowing (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Swallowing (Change from Baseline at Week 52) | 0.00 (1.109) | -0.29 (1.360)
  Memory (Baseline) | 1.56 (1.294) | 1.63 (1.051)
  Memory (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 38
  Memory (Change from Baseline at Week 52) | 0.00 (0.784) | 0.18 (1.218)
  Speech (Baseline) | 1.17 (0.707) | 1.42 (0.722)
  Speech (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Speech (Change from Baseline at Week 52) | 0.14 (0.663) | -0.18 (0.673)
  Eye Movement (Baseline) | 2.11 (0.471) | 1.92 (0.428)
  Eye Movement (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Eye Movement (Change from Baseline at Week 52) | 0.00 (0.679) | -0.06 (0.547)
  Hearing (Baseline): number analyzed (Participants) | 16 | 36
  Hearing (Baseline) | 0.94 (0.998) | 0.94 (1.145)
  Hearing (Change from Baseline at Week 52): number analyzed (Participants) | 9 | 21
  Hearing (Change from Baseline at Week 52) | -0.22 (1.302) | 1.14 (1.236)
  Seizures (Baseline) | 1.00 (1.572) | 1.13 (1.630)
  Seizures (Change from Baseline at Week 52): number analyzed (Participants) | 14 | 34
  Seizures (Change from Baseline at Week 52) | -0.50 (1.286) | -0.06 (0.952)

9. Secondary Outcome: Parts A/B: Change From Baseline to Week 52 in the Total NPC-SS (With Hearing Domain and ABR Modifier Included)
Description: The NPC-SS total score is based on 9 domains including ambulation, fine motor skills, cognition, swallowing, memory, speech, eye movement, hearing (sensorineural) and seizures. A Likert-like scale is used to assign to each domain score of 0 to 5 (better to worse). The total score was the sum of individual components scores which ranges from 0 (best) to 45 (worst), with higher scores indicating more severe clinical impairment.
Time Frame: Baseline, Week 52
Population: mITT population included all randomized participants who received at least one treatment). As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study. Here, overall number of participants analyzed = participants evaluable for this outcome measure, and number analyzed = participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 14 | 25
score on a scale
  Baseline | 15.64 (7.531) | 17.76 (5.349)
  Change from Baseline at Week 52: number analyzed (Participants) | 3 | 4
  Change from Baseline at Week 52 | 0.000 (1.000) | 0.75 (4.500)

10. Secondary Outcome: Parts A/B: Time to One Point Increase (Worsening) in NPC-SS Composite Score
Description: The NPC-SS composite score is the sum of the ambulation, cognition, fine motor, and swallowing domains of the NPC-SS. Each of the four NPC-SS components (ambulation, cognition, fine motor, and swallowing) are rated on a scale from 0 (better) to 5 (worse). The total score was the sum of individual components scores which ranges from 0 (best) to 20 (worst), with higher scores indicating more severe clinical impairment. The product-limit survival analysis method is used to estimate the time to one point increase (worsening) in NPC-SS composite score. Time to worsening in NPC-SS Composite Score defined as the interval from study drug administration to a one point increase in the NPC-SS composite score. If a subject discontinued from the study prior to Week 52, then the subject was censored at time of discontinuation. If a subject completed the Week 52 visit, then the subject was censored at the time of last study visit.
Time Frame: Baseline up to Week 52
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
Days | 118 [55 to 364] | 169 [70 to 278]

11. Secondary Outcome: Parts A/B: Change From Baseline in the Timed Up and Go (TUG) Test at Week 52
Description: The TUG is a test of balance and risk for falls. This test measures the time taken by a participant to walk 3 meters starting from a sitting position and it ends when the participant is seated again.
Time Frame: Baseline, Week 52
Population: mITT population included all randomized participants who received at least one treatment. As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study. Here, overall number of participants analyzed = participants evaluable for this outcome measure, and number analyzed = participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 35
seconds
  Baseline | 18.04 (19.000) | 16.40 (13.218)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 29
  Change from Baseline at Week 52 | 0.86 (19.232) | 2.70 (9.633)

12. Secondary Outcome: Parts A/B: Change From Baseline in the 9-Hole Peg Test at Week 52
Description: The 9-Hole Peg Test is a brief, standardized, quantitative test of upper extremity function. The participant picks up 9 pegs puts them in a block containing nine empty holes, and, once they are in the holes, removes them again as quickly as possible one at a time. The total time to complete the task is recorded.
Time Frame: Baseline, Week 52
Population: mITT population included all randomized participants who received at least one treatment (sham or adrabetadex). As per planned analysis, efficacy data were collected and presented by overall randomized treatment assignment (either sham or adrabetadex). These two treatment arms (either sham or adrabetadex) combine data from Parts A and B of the study. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 18 | 38
seconds | -1.49 (15.958) | -1.79 (34.760)

13. Secondary Outcome: Parts A/B: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an adverse event (AE) with onset on or after start of study Drug. An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 52
Population: Safety population was defined as all randomized participants who received at least 1 procedure (adrabetadex infusion via LP or sham).
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Adrabetadex 900 mg: Participants received 4 lumbar IT infusions of adrabetadex 900 mg once every 2 weeks.
Arm/Group | Part A: Adrabetadex 900 mg | Part A: Adrabetadex 1200 mg | Part A: Adrabetadex 1800 mg | Part A: Sham Control | Part B: Adrabetadex 900 mg | Part B: Sham Control
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 29 | 15
Participants | 3 | 3 | 3 | 3 | 28 | 14

14. Secondary Outcome: Parts A/B: Change From Baseline to Week 52 in Mean Annualized Rate of Change (Slope) of NPC-SS Composite Score
Description: The NPC-SS composite score is the sum of the ambulation, cognition, fine motor, and swallowing domains of the NPC-SS. Each of the four NPC-SS components (ambulation, cognition, fine motor, and swallowing) are rated on a scale from 0 (better) to 5 (worse). The total score was the sum of individual components scores which ranges from 0 (best) to 20 (worst), with higher scores indicating more severe clinical impairment. The Annualized rate of change (Slope) is calculated as 365.25 *([measurement at post-baseline visit - measurement at baseline]/[date of post-baseline visit - date of baseline visit + 1]).
Time Frame: Baseline, Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on NPC-SS scale/year
Arm/Group | Sham Control | Adrabetadex
Number analyzed (Participants) | 14 | 34
score on NPC-SS scale/year | -0.05 (1.640) | 0.08 (2.441)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Safety population was defined as all randomized participants who received at least 1 procedure (adrabetadex infusion via LP or sham).
Arm/Group | Part A: Adrabetadex 900 mg | Part A: Adrabetadex 1200 mg | Part A: Adrabetadex 1800 mg | Part A: Sham Control | Part B: Adrabetadex 900 mg | Part B: Sham Control
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 0/29 | 1/15
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 0/3 | 16/29 | 3/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 28/29 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Adrabetadex 900 mg (N=3) | Part A: Adrabetadex 1200 mg (N=3) | Part A: Adrabetadex 1800 mg (N=3) | Part A: Sham Control (N=3) | Part B: Adrabetadex 900 mg (N=29) | Part B: Sham Control (N=15)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 3 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hearing Impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 3 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Abasia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Croup Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Stoma Site Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Postictal Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1
Speech Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mutism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 0
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Adrabetadex 900 mg (N=3) | Part A: Adrabetadex 1200 mg (N=3) | Part A: Adrabetadex 1800 mg (N=3) | Part A: Sham Control (N=3) | Part B: Adrabetadex 900 mg (N=29) | Part B: Sham Control (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (13) | 1 (2)
Dysacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing Impaired (Ear and labyrinth disorders) | 2 (4) | 1 (5) | 1 (4) | 0 (0) | 8 (18) | 6 (11)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 2 (5) | 1 (2) | 0 (0) | 10 (27) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (11) | 0 (0)
Early Menarche (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid Haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 9 (16) | 1 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (7) | 4 (7)
Faecal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (4)
Faeces Discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malpositioned Teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (5) | 2 (3) | 1 (1) | 8 (19) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (6) | 3 (3) | 1 (3) | 0 (0) | 15 (35) | 2 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (14) | 1 (1)
Facial Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (8) | 2 (4) | 2 (7) | 1 (2) | 12 (29) | 2 (3)
Gait Disturbance (General disorders) | 1 (3) | 1 (2) | 3 (10) | 0 (0) | 11 (47) | 2 (6)
Injection Site Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 12 (23) | 3 (7)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Acute Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 3 (7) | 3 (4)
Tinea Manuum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (9)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (19) | 2 (4)
Eye Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (63) | 1 (10)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural Headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 1 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1)
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tympanometry Abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Feeding Disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (6) | 2 (7) | 1 (5) | 2 (3) | 14 (68) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (1) | 1 (1) | 0 (0) | 3 (9) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 5 (14) | 1 (2)
Altered State Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 1 (3) | 1 (2) | 3 (11) | 0 (0) | 7 (34) | 2 (4)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Cataplexy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (14) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Fine Motor Skill Dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (9) | 1 (1) | 9 (65) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyporesponsive To Stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Language Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 1 (2)
Motor Dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 1 (1)
Somnolence (Nervous system disorders) | 1 (3) | 1 (3) | 2 (3) | 1 (1) | 3 (33) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Viith Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 2 (6) | 1 (2)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased Eye Contact (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emotional Distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Personality Change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staring (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Stereotypy (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 6 (13) | 4 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (20) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (30)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT02534844/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT02534844/SAP_001.pdf